CLINICAL TRIAL: NCT05002595
Title: Comparison of Helicobacter Pylori Treatment Between Modified Quadruple Therapy and Tailored Eradication Based on the Presence of Clarithromycin Resistance
Brief Title: H. Pylori Treatment Between Modified Quadruple Regimen and Tailored Therapy
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Associate Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2021
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen would be obtained for urease test (commercial name: CLOtest) or molecular test (DPO-PCR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modified quadruple therapy: pantoprazole 40mg bid, amoxicillin 1000mg bid, metronidazole 750mg bid, bismuth subcitrate 600mg bid for 14 days
  Interventions: Drug: H. pylori eradication
- Tailored eradication: pantoprazole 40mg bid, amoxicillin 1000mg bid, clarithromycin 500mg bid or pantoprazole 40mg bid, tetracycline 1000mg bid, metronidazole 750mg bid, bismuth subcitrate 600mg bid for 7 days
  Interventions: Drug: H. pylori eradication

INTERVENTIONS:
Drug: H. pylori eradication — Antimicrobial agents for H. pylori eradication

SUMMARY:
The rate of H. pylori resistance to antimicrobial agents including clarithromycin (CAM) has increased worldwide. Eradication failure using triple therapy is strongly associated with CAM-resistant H. pylori. The tailored therapy is defined as a targeted H. pylori eradication which emphasizes on predicting individual drug responses before treatment.

Dual priming oligonucleotide (DPO)-based multiplex polymerase chain reaction (PCR) was developed to diagnose H. pylori infection and identify CAM resistance. The use of DPO-PCR has increased the tailored H. pylori eradication rate in Korea. If DPO-PCR testing is not available, a 14-day modified bismuth-containing quadruple regimen is recommended as a first-line H. pylori eradication. However, there is no comparison study between modified quadruple therapy and tailored eradication based on the presence of CAM resistance using DPO-PCR.

DETAILED DESCRIPTION:
The investigators aim to evaluate the success rate, adverse drug events, and cost-effectiveness of modified quadruple therapy, compared with tailored eradication based on the presence of CAM resistance.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected patients
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
H. pylori infection status | 6 weeks
  Rate of successful H. pylori eradication

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JH, Jin SY, Park S. Comparison of tailored Helicobacter pylori eradication versus modified bismuth quadruple therapy in Korea: a randomized controlled trial. Expert Rev Anti Infect Ther. 2022 Jun;20(6):923-929. doi: 10.1080/14787210.2022.2017280. Epub 2021 Dec 20. PMID 34883037